CLINICAL TRIAL: NCT03213769
Title: Clinical Evaluation of Topical Coenzyme Q10 in Management of Oral Aphthous Ulcer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mostafa Abdelsamie Bakry Nafie, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1990
Record Dates: First submitted 2017-07-05; First posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Oral Aphthous Ulcer
Keywords: oral minor aphthous ulcer; topical Q10 gel; topical antioxidant; oral recurrent aphthous ulcer; oral aphthous stomatitis
MeSH Terms: conditions — Foot-and-Mouth Disease

STUDY DESIGN:
Intervention Model Description: controlled randimized clinical trial
Who Masked: Participant, Investigator
Masking Description: double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- topical coenzyme Q10 gel (Active Comparator): Q10 gel will give 2 times /day after breakfast and evening meal for 7 days.
  Interventions: Drug: topical coenzyme Q10 gel
- carbapol gel (Placebo Comparator): placebo carbapol gel will give 2 times /day after breakfast and evening meal for 7 days.
  Interventions: Drug: Carpabol gel

INTERVENTIONS:
Drug: topical coenzyme Q10 gel — Q10 gel will give 2 times /day after breakfast and evening meal for 7 days.
  Arms: topical coenzyme Q10 gel
Drug: Carpabol gel — placebo carbapol gel will give 2 times /day after breakfast and evening meal for 7 days.
  Arms: carbapol gel

SUMMARY:
Recurrent oral aphthous ulcer is the most common oral lesion in occurrence and one of cause is oxidative stress so investigators need to use antioxidant drugs like topical coenzyme Q10 gel to treat the lesion and more safe for the participants.

DETAILED DESCRIPTION:
Double randomized clinical trial study using two parallel group suffer from oral aphthous ulcer one take antioxidant topical q10gel and other group take placebo carpabol gel two times per day for seven days measuring outcome at fourth and seventh day including pain; healing period and clinical parameters.

Sample size of study include 26 in each group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with free medical history and no systemic diseases16.
* Patients clinically diagnosed as suffering from symptomatic oral minor aphthous ulcers.
* Patients who agreed to take medications.

Exclusion Criteria:

* Patients suffering from any systemic disease as Crohn's disease, Behcet's disease and others.
* Anemic and leukemic patients (using complete blood count investigation)
* Patients taking systemic drugs such as systemic steroids and other immunosuppressive therapy.
* Patients treated with any oral topical medications 48h before the study27.
* Pregnant and lactating mothers.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2017-07 (Estimated); Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
visual analogue scale | 7 days
  pain

SECONDARY OUTCOMES:
scoring system(0-3) | 7 days
  Erythema surround lesion
cross sectional area William periodontal probe/mm | 7 days
  Cross sectional area

CONTACTS AND LOCATIONS:
Overall Officials: fatheya zahran, professor, Study Director — faculty of dentistry -CairoU

REFERENCES:
- [Background] Sawair FA. Recurrent aphthous stomatitis: do we know what patients are using to treat the ulcers? J Altern Complement Med. 2010 Jun;16(6):651-5. doi: 10.1089/acm.2009.0555. PMID 20569032
- [Background] Scully C, Felix DH. Oral medicine--update for the dental practitioner. Aphthous and other common ulcers. Br Dent J. 2005 Sep 10;199(5):259-64. doi: 10.1038/sj.bdj.4812649. PMID 16155535
- [Background] Momen-Beitollahi J, Mansourian A, Momen-Heravi F, Amanlou M, Obradov S, Sahebjamee M. Assessment of salivary and serum antioxidant status in patients with recurrent aphthous stomatitis. Med Oral Patol Oral Cir Bucal. 2010 Jul 1;15(4):e557-61. doi: 10.4317/medoral.15.e557. PMID 20173724
- [Background] Littarru GP, Tiano L. Bioenergetic and antioxidant properties of coenzyme Q10: recent developments. Mol Biotechnol. 2007 Sep;37(1):31-7. doi: 10.1007/s12033-007-0052-y. PMID 17914161
- [Background] Tarakji B, Gazal G, Al-Maweri SA, Azzeghaiby SN, Alaizari N. Guideline for the diagnosis and treatment of recurrent aphthous stomatitis for dental practitioners. J Int Oral Health. 2015 May;7(5):74-80. PMID 26028911
- [Background] Prakash S, Sunitha J, Hans M. Role of coenzyme Q(10) as an antioxidant and bioenergizer in periodontal diseases. Indian J Pharmacol. 2010 Dec;42(6):334-7. doi: 10.4103/0253-7613.71884. PMID 21189900
- [Background] Preeti L, Magesh K, Rajkumar K, Karthik R. Recurrent aphthous stomatitis. J Oral Maxillofac Pathol. 2011 Sep;15(3):252-6. doi: 10.4103/0973-029X.86669. PMID 22144824
- [Background] Hamdy AA, Ibrahem MA. Management of aphthous ulceration with topical quercetin: a randomized clinical trial. J Contemp Dent Pract. 2010 Jul 1;11(4):E009-16. PMID 20953559